CLINICAL TRIAL: NCT06898047
Title: CORRELATE-UK: COnsistency of Response With RimegEpant Oral Lyophilisate in Acute Treatment of migrainE in the United Kingdom
Brief Title: Consistency of Response With Rimegepant in Acute Treatment of Migraine
Acronym: CORRELATE-UK
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4951071; CORRELATE-UK (Other: Alias Study Number)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; Acute migraine treatment; rimegepant
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Rimegepant users: Participants with current prescription of rimegepant for acute treatment of migraine
  Interventions: Drug: Rimegepant for acute migraine treatment

INTERVENTIONS:
Drug: Rimegepant for acute migraine treatment — Rimegepant for acute migraine treatment

SUMMARY:
This is a non-interventional, prospective study that will enroll participants with migraine in the United Kingdom currently in use of rimegepant to acutely treat migraine attacks. Participants will be followed up for up to 12 weeks and will complete a daily questionnaire to self-report the consistency of response to rimegepant in acute treatment of migraine.

DETAILED DESCRIPTION:
This is a prospective observational, real-world cohort study of the patient-reported consistency of response to rimegepant in acute treatment of migraine. Longitudinal data capture will allow the determination of treatment effectiveness across multiple attacks, while the observational design will ensure the data reflect a real-world setting. In addition, a patient-centered real-time approach will allow for capture of granular data and will minimize patient recall bias, which is important for subjective outcomes such as pain. Patient reported outcome measures will be collected at study enrolment, daily during the 12-week observation period, and at the end of the study period.

The study will be conducted in the United Kingdom (UK). Potential participants will be identified and selected from UK healthcare institutions. Both patients diagnosed with episodic and chronic migraine will be included, with a split of approximately 50% of each group. Participants will be enrolled into the study over a period of approximately 6 months. The total data collection period will be approximately 9 months. Potentially eligible patients will receive briefing materials during a routine in-person consultation, or via email. Interested patients will use a link and a unique ID and PIN to complete a study eligibility screener within the study web application. The screener will consist of a series of demographic and clinical history questions. Participants who successfully complete the eligibility will then be able to proceed to the consent stage. Informed consent will also be provided within the study web application.

Consented participants will be required to complete a series of baseline demographic and clinical questions within a window of 72h from registration. A completion reminder will be sent every 24h until the completion window closes. Each participant will be followed up for 12 weeks. During this period, participants will receive an SMS with a link to the study website at the same time every day. A single click on the phone will take participants to the daily migraine survey. Two custom questions asking about migraine symptom occurrence and rimegepant use in the previous 24h will be presented to every participant daily from Day 1 to Day 84. A series of custom follow-up questions, asking further information about any migraine symptoms and related treatment, will be presented based on participant responses to questions 1 and 2 . A completion window of four days (96h) will be allowed for the daily questions. In case participants are still experiencing some migraine symptoms when prompted, they will be able to save their responses and return at a later time within the completion window. On Days 0, 28, 56 and 84 of follow-up, a menstruation question will be presented to all participants. At the end of the 12-week follow-up, the mTOQ-6 Likert version and the TSQM-II questionnaire will be presented to all participants.

ELIGIBILITY:
Inclusion criteria

1. UK resident.
2. At least 18 years of age.
3. Migraine diagnosis confirmed by healthcare professional.
4. Current prescription of rimegepant for acute treatment of migraine.
5. Experienced at least 4 migraine attacks per month prior to study enrolment.
6. In the case of participants receiving preventive migraine treatment:

   * For oral preventives, the treatment must be "stable" i.e., final dosing regimen has been found.
   * For migraine preventives administered monthly, the participant must have had their most recent treatment within the 3 weeks prior to study enrolment.
   * For migraine preventives administered quarterly, the participant must have had their most recent treatment within the 2 months prior to study enrolment.
   * If the last treatment is not within the stipulated period, participants will be asked to provide the date of the next scheduled treatment, after which the participant may be invited back to enrol into the study.
7. Evidence of a personally signed (or acknowledged if obtained electronically or online) and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.

Exclusion criteria

1. Current use of rimegepant as a preventive migraine medication.
2. Current diagnosis of any of the following conditions:

   * new daily persistent headache
   * chronic daily headache
   * cluster headache
   * post-traumatic headache
   * hemicrania continua
   * major depression
   * pain syndromes other than migraine (e.g. fibromyalgia)
   * psychiatric conditions (e.g., schizophrenia)
   * dementia
   * significant neurological disorders other than migraine.
3. Current prescription of any of the following medications:

   * Strong inhibitors of CYP3A4
   * Strong or moderate inducers of CYP3A4
4. Patients participating in a migraine-related clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants living in the United Kingdom, with a migraine diagnosis confirmed by a healthcare professional, experiencing at least 4 migraine attacks per month, with a current prescription of rimegepant for acute treatment of migraine, and, if receving preventive migraine treatment, must be stable before enrollment. Participants will be excluded if they are currently using rimegepant as preventive migraine treatment, if present other specific neurological conditions, if currently prescribed with drugs that may indude or inhibits CYP3A4, or if they are participating in a migraine-related clinical trial. All participants enrolled must acknowledge their participation in the study informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to Meaninful Pain Relief (MPR) post-dosing | Daily (within 24hs post dose)
  Proportion of participants who report MPR: within 1 hour post dose; 1-2 hours post dose; Over 2 hours up to 4 hours post dose; More than 4 hours post dose; who have not achieved MPR and took the medication more than 2 hours before completing the survey; who have not achieved MPR and took the medication less than 2 hours before completing the survey

SECONDARY OUTCOMES:
Time to improvement in non-pain symptoms post-dosing | Daily (within 24hs post dose)
  Proportion of participants who report improvement in any non-pain symptoms: within 1 hour post dose; 1-2 hours post dose; Over 2 hours up to 4 hours post dose; More than 4 hours post dose; who have not had a meaninful improvement and took the medication more than 2 hours before completing the survey; who have not had a meaninful improvement and took the medication less than 2 hours before completing the survey.
Acute migraine treatment optmization | 12 weeks follow up
  Proportion of participants on an acute treatment regimen over a 12-week follow up period.
Acute migraine treatment optmization | 12 weeks follow up
  Description of the acute migraine treatments used over a 12-week follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951071